CLINICAL TRIAL: NCT03785704
Title: Clinical Study of Xinmailong Injection on Reducing Cardiovascular Toxicity in Adjuvant Chemotherapy in Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Fei Ma, Deputy director of oncology, Peking Union Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC1786
Record Dates: First submitted 2018-12-05; First posted 2018-12-24 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Breast Neoplasms; Cardiac Event; Chemotherapeutic Toxicity
Keywords: Xinmailong injection; anthracycline induced cardiac toxicity
MeSH Terms: conditions — Breast Neoplasms; Cardiovascular Diseases | interventions — xinmailong

STUDY DESIGN:
Intervention Model Description: Totally 60 subjects will be included in the study.Random assignment was 1:1 to Xinmailong injection group and control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xinmailong injection group (Experimental): given 5 mg/kg of Xinmailong injection every cycle on d0, d1, d2, d3, d4 on the same chemotherapy regimen (EC-T) as those in the control group.
  Interventions: Drug: Xinmailong Injection
- control group (No Intervention): receive conventional EC-T regimen chemotherapy (Epirubicin 45mg/m2 d1, 2 + cyclophosphamide 600mg/ m2 d1, repeated every 14 or 21 days for 4 cycles, followed by paclitaxel 175 mg/m2 (or docetaxel 75 mg/m2) on day 1, repeated every 21 days for 4 cycles).

INTERVENTIONS:
Drug: Xinmailong Injection — Xinmailong injection is extracted, separated, purified and refined from Periplaneta americana. It is the second class of new drugs and the only small molecular bioactive peptide preparation approved by the State Pharmaceutical Administration (P.R.China) for the prevention and treatment of heart failure. Its main constituents include complex nucleoside bases and binding amino acids.
  Arms: Xinmailong injection group

SUMMARY:
Totally 60 subjects will be included in the study. The present study was aimed to observe and evaluate the effect of Xinmailong injection on reducing cardiovascular toxicity associated with adjuvant chemotherapy after breast cancer surgery. The primary endpoint was 6 months of cardiac safety. Secondary endpoints included 3 months of cardiac safety, adverse events (AE), severe adverse events (SAE), and DFS.

DETAILED DESCRIPTION:
After signing the informed consent, the patients in the control group will receive Epirubicin 45mg/m2 d1, 2 + cyclophosphamide 600mg/ m2 d1, repeated every 14 or 21 days for 4 cycles, followed by paclitaxel 175 mg/m2 (or docetaxel 75 mg/m2) on day 1, repeated every 21 days for 4 cycles. Patients in the Xinmailong group were given 5 mg/kg of Xinmailong injection every cycle on d0, d1, d2, d3, d4 on the same chemotherapy regimen as those in the control group. The patients-general condition, vital signs, blood routine, liver and kidney function, electrocardiogram, myocardial enzymes, troponin, BNP and echocardiography should be examined every week. Breast ultrasound were performed every week. Chest CT were evaluated after 8 cycles of chemotherapy.

After adjuvant chemotherapy, adjuvant radiotherapy and endocrine therapy were given according to the situation, and long-term survival was observed.

The patients will be followed up for 5 years, once every 6 months with in 1-3 years, once every 12 months within 4-5 years.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years, female;
2. after radical mastectomy, EC - T adjuvant chemotherapy is planned.
3. No relevant treatment (such as antineoplastic therapy, immunotherapy, etc.) that may affect the outcome of treatment was received before admission.
4. ECOG PS score: 0-2 points;
5. Laboratory criteria:

   * white blood cells were more than 4 x 109 /L, and neutrophil count (ANC) was more than 1.5 x 109 /L.

     * platelet (>100 *109/L); hemoglobin (>10g/dL); serum creatinine (<1.5 *normal value) upper limit (ULN); aspartate aminotransferase (AST) (<2.5 *ULN); alanine aminotransferase (ALT) (<2.5 *ULN); total bilirubin (<1.5 *ULN); serum creatinine (<1.5 *ULN); the volunteers voluntarily joined the study, signed informed consent, and had good compliance and follow-up.

Exclusion Criteria:

1. cockroach or xinmailong allergy (including xinmailong test positive).
2. Pregnant or lactation woman
3. severe bleeding tendency;
4. With mental disease
5. With severe infection or active gastrointestinal ulcers
6. allergic to chemotherapeutic agents;
7. Disease-free period of other malignant tumor is less than 5 years(except cured basal cell skin cancer and cervical carcinoma in situ).
8. With severe liver disease (such as cirrhosis), kidney disease, respiratory disease or diabetes
9. taking part or participating in other clinical trials within one month.
10. previous history of severe cardiovascular disease or cardiovascular disease risk factors were ≥ 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
The rate of no cardiac events during chemotherapy | up to 12 months
  Adverse events (AEs) and laboratory tests graded according to the NCI CTCAE (version 4.0) .No cardiac events were defined until all relevant indicators (Electrocardiograph, Echcardiography and myocardial enzyme) were normal during chemotherapy.

SECONDARY OUTCOMES:
Disease-free survival (DFS) | 5 years
  The time between the start of a randomized clinical trial and the onset of disease recurrence or death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Beijing, China